CLINICAL TRIAL: NCT07149714
Title: Temporary Mechanical Circulatory Support With the iVAC 2L Transaortic Device in High-risk Percutaneous Coronary Intervention
Brief Title: Temporary MCS With the iVAC 2L Transaortic Device in High-risk PCI
Acronym: POTOK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Principal Investigator, Dmitry Pevzner, Head of the Emergency Cardiology Department, National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-32-1
Record Dates: First submitted 2025-08-13; First posted 2025-09-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Cardiovascular Disease; Multivessel Coronary Artery Disease; Coronary Artery Disease; Cardiogenic Shock; Acute Heart Failure (AHF); Chronic Heart Failure; Percutaneous Coronary Intervention
Keywords: Mechanical circulatory support; High-Risk Percutaneous Coronary Intervention; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Shock, Cardiogenic

STUDY DESIGN:
Intervention Model Description: 100 pts with coronary artery disease with indications for High-Risk Percutaneous Coronary Intervention and no contradictions for the placement of the iVAC2L will be enrolled. The risk of PCI will be assessed by the institution's heart team (presence of severe coronary artery disease, acute coronary syndrome, other comorbidities including renal disease, diabetes mellitus, chronic and acute heart failure etc.). Pts participating in the clinical trial are expected to remain hospitalized for approximately 7-14 days and will be followed for 360 days (with an acceptable range of 350-370 days) after the intervention or until the occurrence of the primary endpoint.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safety and clinical efficacy of temporary MCS with the iVAC 2L transaortic device in high-risk PCI (Experimental): 100 pts with coronary artery disease with indications for High-Risk Percutaneous Coronary Intervention and no contradictions for the placement of the iVAC2L.
  Interventions: Device: iVAC 2L

INTERVENTIONS:
Device: iVAC 2L — The goal of this study is to investigate the safety and clinical efficacy of temporary mechanical support system with the iVAC 2L transaortic device in high-risk percutaneous coronary intervention (PCI) in Russia and Belarus. The POTOK trial will include patients with indications for elective, urgent and emergency PCI.

SUMMARY:
Patients with coronary artery disease and undergoing high-risk percutaneous coronary intervention (PCI) are at increased risk of hemodynamic instability and poor outcomes. Mechanical circulatory support (MCS) devices may offer hemodynamic stabilization during PCI, potentially improving short- and long-term outcomes. The study rationale is to investigate the safety and clinical efficacy of temporary MCS with the iVAC 2L transaortic device in high-risk percutaneous coronary intervention.

The transaortic system for short-term circulatory support with pulsatile blood flow iVAC 2L consists of an external membrane pump, a 17Fr diameter catheter for reversed blood flow (intake cannula) with a patented two-way rotary valve.

The pump has two chambers, one for blood and one for helium, separated by a flexible diaphragm. The blood chamber connects to the catheter and the air chamber connects to a standard IABP console. The bi-directional valve is located 72 mm from the aspiration tip of the catheter and determines the direction of blood flow. The catheter is advanced retrogradely through the common femoral artery so that the tip is located in the left ventricular (LV) cavity and the valve is in the ascending aorta. Synchronized with the cardiac cycle via ECG, the device draws blood from the LV into the pump chamber during systole and ejects blood from the pump into the ascending aorta during diastole.

The primary composite outcome is all-cause mortality, including acute myocardial infarction, stroke and TIA during hospitalization and at Day 360 of follow-up, expressed as a percentage of total patients.

DETAILED DESCRIPTION:
Although coronary artery bypass grafting (CABG) remains the standard treatment for patients with multivessel coronary artery disease, there is growing interest in performing protected percutaneous coronary intervention (PCI) in high-risk patients. Protected PCI involves the use of temporary mechanical circulatory support (MCS) devices during and shortly after the procedure to maintain hemodynamic stability and reduce the risk of complications such as acute left ventricular failure. This approach offers a safer alternative to open-heart surgery in patients for whom CABG poses significant operative risks. The study rationale is to investigate the safety and clinical efficacy of temporary MCS with the iVAC 2L transaortic device in high-risk percutaneous coronary intervention.

On admission patients will undergo ECG, echocardiography, routine blood tests including complete blood count and basic metabolic panel. After then the patient's risk will be assessed by the institution's heart team (presence of severe coronary artery disease, acute coronary syndrome, other comorbidities including renal disease, diabetes mellitus, chronic and acute heart failure etc.).

For placement of the iVAC 2L transaortic device the patient will be transported to the X-ray operating room. The transaortic system for short-term circulatory support with pulsatile blood flow that consists of three main components: an external membrane pump, a 17Fr diameter catheter for reversed blood flow (intake cannula) and a patented two-way rotary valve. The pump has two chambers, one for blood and one for helium, separated by a flexible diaphragm. The blood chamber connects to the catheter and the air chamber connects to a standard IABP console. The bi-directional valve is located 72 mm from the aspiration tip of the catheter and determines the direction of blood flow. The catheter is advanced retrogradely through the common femoral artery so that the tip is located in the left ventricular (LV) cavity and the valve is in the ascending aorta. Synchronized with the cardiac cycle via ECG, the device draws blood from the LV into the pump chamber during systole and ejects blood from the pump into the ascending aorta during diastole. Advantages of the iVAC 2L include a minimally invasive implantation technique, pulsatile flow that may be more physiologic compared to continuous flow devices, and a lower risk of hemolysis and vascular complications compared to other MCS devices.

After surgery further monitoring of the patient will be carried out in the intensive care unit. During hospitalization treatment and diagnostic evaluation of patients will be done according to current clinical practice guidelines.

The primary composite outcome is all-cause mortality, including acute myocardial infarction, stroke and TIA during hospitalization and at Day 360 of follow-up, expressed as a percentage of total patients.

ELIGIBILITY:
Inclusion Criteria:

* Multidisciplinary heart team consensus for high-risk PCI. HR-PCI was defined as any percutaneous intervention for coronary disease involving an unusually high risk of periprocedural circulatory collapse.
* Signed Informed Consent to participate in the study

Exclusion Criteria:

* Femoral artery diameter < 6.0mm
* Significant biventricular or right heart failure
* Thrombus in the left ventricle
* Presence of a mechanical aortic valve
* Aortic valve stenosis/calcification (equivalent to an orifice area of 0.6 cm2 or less) or moderate-to-severe aortic insufficiency (echocardiographic assessment graded as ≥+2)
* Severe peripheral arterial disease precluding placement of the iVAC2L
* Combined cardiorespiratory failure
* Presence of an atrial or ventricular septal defect (including post infarct VSD)
* Left ventricular rupture
* Cardiac tamponade
* Presence of any other subtype of shock
* Known severe comorbidities independently affecting prognosis (chronic renal or liver failure, active malignancies etc.)
* Recent major bleeding event (< 3 months)
* Recent stroke (< 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2028-02-17 (Estimated); Study Completion 2029-02-17 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | At day 7 after PCI or at discharge, if earlier. At day 360 of follow-up.
  Constitutes one of the components of the MACCE composite endpoint: all-cause mortality, acute myocardial infarction, stroke or transient ischemic attack (TIA), and repeat revascularization (PCI or CABG).

SECONDARY OUTCOMES:
Major vascular complications | From the beginning of the PCI until its conclusion, the PCI is estimated to be from 40 to 270 minutes.
  Complications include development of limb ischemia after PCI, bleeding in access site, development of arteriovenous fistula and infectious access site complications, as per VARC-2 definitions.
Incidence of recurrent myocardial infarction or reinfarction | During the 360-day follow-up period
  According to the Fourth Universal Definition of Myocardial Infarction (ESC, 2018)
Angiographic failure | Immediately after PCI.
  Angiographic failure/procedural failure, as defined in the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention Circulation: post-procedure TIMI flow < grade III, residual stenosis (>50% post-balloon or > 10% post stenting), or presence of thrombus, side branch loss or flow limiting dissection. It is a binary outcome (yes/no answer).
Incidence of intraprocedural complications | From the beginning of the PCI until its conclusion, the PCI is estimated to be from 40 to 270 minutes.
  Including life-threatening ventricular arrhythmias, cardiac arrest, and progression of cardiogenic shock (as per SCAI classification)
Left ventricular myocardial function | At day 7 after PCI or at discharge, if earlier.
  Ejection fraction, measured in percentages; based on trans-thoracic echocardiographic assessment
Incidence of acute kidney injury | At day 7 after PCI or at discharge, if earlier.
  Assessed via changes in serum creatinine and/or urine output, according to KDIGO 2012 criteria
Angiographic characteristics | From the beginning of the PCI until its conclusion. The PCI is estimated to be from 40 to 270 minutes.
  SYNTAX score (to estimate the complexity of coronary artery disease, higher score is associated with poor clinical outcomes) before and after the procedure, anatomical characteristics of the coronary arteries (three-vessel, unprotected left main, last remaining vessel and bifurcational lesions), the use of intravascular imaging (ex. IVUS).
Number of Participants with ventricular arrhythmias | From the beginning of the PCI until its conclusion, the PCI is estimated to be from 40 to 270 minutes. At day 7 after PCI or at discharge, if earlier.
  VT requiring cardioversion and/or need for CPR. Binary outcome, VF during hospitalization.
Number of participants with progression of cardiogenic shock | From the beginning of the PCI until its conclusion, the PCI is estimated to be from 40 to 270 minutes. At day 7 after PCI or at discharge, if earlier.
  As defined by SCAI-CSWG in 2022
Number of participants with major bleeding | At day 7 after PCI or at discharge, if earlier.
  Major bleeding (BARC 3 to 5) after PCI, according to the BARC Bleeding Classification 2011.
Number of participants with acute myocardial infarction | At day 7 after PCI or at discharge, if earlier. At day 360 of follow-up.
  According to the Fourth Universal Definition of Acute Myocardial Infarction (ESC, 2018). Constitutes one of the components of the MACCE composite endpoint: all-cause mortality, acute myocardial infarction, stroke or transient ischemic attack (TIA), and repeat revascularization (PCI or CABG).
Number of participants with stroke or transient ischemic attack | At day 7 after PCI or at discharge, if earlier. At day 360 of follow-up.
  As per VARC 2 definitions 2013. Constitutes one of the components of the MACCE composite endpoint: all-cause mortality, acute myocardial infarction, stroke or transient ischemic attack (TIA), and repeat revascularization (PCI or CABG).
Repeat revascularization | At day 7 after PCI or at discharge, if earlier. At day 360 of follow-up.
  As per ARC definition 2007. Constitutes one of the components of the MACCE composite endpoint: all-cause mortality, acute myocardial infarction, stroke or transient ischemic attack (TIA), and repeat revascularization (PCI or CABG).
Intraprocedual device-related characteristics | From the beginning of the PCI until its conclusion, the PCI is estimated to be from 40 to 270 minutes.
  Implantation failure, device operating mode (internal or ECG synchronized), duration of device runtime (measured in minutes), device dislocation, use of other MCS
Change in Left ventricular ejection fraction | From baseline (before the PCI) to the moment of discharge, typically on the 5-7 day after PCI.
  Numerical continuous variable. Change in LVEF measured by trans-thoracic echocardiography at baseline and discharge. Measured in percentages.
Severity of aortic valve regurgitation | At baseline (before the PCI).
  Based on trans-thoracic echocardiographic assessment as per European Association of Echocardiography guidelines.
Severity of mitral valve stenosis | At baseline (before the PCI).
  Based on trans-thoracic echocardiographic assessment as per European Association of Echocardiography guidelines.
Severity of triscupid valve regurgitation | At baseline (before the PCI).
  Based on trans-thoracic echocardiographic assessment as per European Association of Echocardiography guidelines.
Severity of aortic valve stenosis | At baseline (before the PCI).
  Based on trans-thoracic echocardiographic assessment as per European Association of Echocardiography guidelines.
Severity of mitral valve regurgitation | At baseline (before the PCI).
  Based on trans-thoracic echocardiographic assessment as per European Association of Echocardiography guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Pevzner, MD, Principal Investigator — National Medical Research Center for Cardiology, Ministry of Health of Russian Federation; Evgeniy Merkulov, MD, Principal Investigator — National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Locations (1):
- NMRCCardiologyRu, Moscow, Russia

REFERENCES:
- [Background] Bulum J, Bastos MB, Hlinomaz O, Malkin O, Pawlowski T, Dragula M, Gil R. Pulsatile Left Ventricular Assistance in High-Risk Percutaneous Coronary Interventions: Short-Term Outcomes. J Clin Med. 2024 Sep 10;13(18):5357. doi: 10.3390/jcm13185357. PMID 39336843
- [Background] Samol A, Wiemer M, Kaese S. Comparison of a pulsatile and a continuous flow left ventricular assist device in high-risk PCI. Int J Cardiol. 2022 Aug 1;360:7-12. doi: 10.1016/j.ijcard.2022.05.038. Epub 2022 May 18. PMID 35597491
- [Background] Ameloot K, B Bastos M, Daemen J, Schreuder J, Boersma E, Zijlstra F, Van Mieghem NM. New-generation mechanical circulatory support during high-risk PCI: a cross-sectional analysis. EuroIntervention. 2019 Aug 29;15(5):427-433. doi: 10.4244/EIJ-D-18-01126. PMID 30741638
- [Background] Bastos MB, van Wiechen MP, Van Mieghem NM. PulseCath iVAC2L: next-generation pulsatile mechanical circulatory support. Future Cardiol. 2020 Mar;16(2):103-112. doi: 10.2217/fca-2019-0060. Epub 2020 Jan 14. PMID 31934785
- [Background] den Uil CA, Daemen J, Lenzen MJ, Maugenest AM, Joziasse L, van Geuns RJ, Van Mieghem NM. Pulsatile iVAC 2L circulatory support in high-risk percutaneous coronary intervention. EuroIntervention. 2017 Feb 20;12(14):1689-1696. doi: 10.4244/EIJ-D-16-00371. PMID 28216471
- [Background] Bastos MB, McConkey H, Malkin O, den Uil C, Daemen J, Patterson T, Wolff Q, Kardys I, Schreuder J, Lenzen M, Zijlstra F, Redwood S, Van Mieghem NM. Effect of Next Generation Pulsatile Mechanical Circulatory Support on Cardiac Mechanics: The PULSE Trial. Cardiovasc Revasc Med. 2022 Sep;42:133-142. doi: 10.1016/j.carrev.2022.03.013. Epub 2022 Mar 14. PMID 35331637